CLINICAL TRIAL: NCT06856928
Title: Impact of Antiobesity Medications on Appetite and Appetite-related Hormones and Metabolites.
Status: Not yet recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Mark Ezpeleta, Post Doctoral Fellow, University of Colorado, Denver
Other Study IDs: 24-1896
Record Dates: First submitted 2025-02-13; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Drug
Keywords: appetite-related hormones; appetite; metabolites
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Early Group: Participants in the early group are individuals that have established agreements with their clinical providers to begin treatment with semaglutide or tirzepatide as part of their ongoing weight management strategy.
  These participants will complete a meal challenge before they start the medication and 6 weeks after starting medication.
  Interventions: Other: Meal Challenge
- Late Group: Participants in the late group are individuals that have lost >12% of their body weight on either semaglutide or tirzepatide and are still taking the medication.
  These participants will complete a meal challenge before they discontinue medication and 3 weeks after discontinuing the medication.
  Interventions: Other: Meal Challenge

INTERVENTIONS:
Other: Meal Challenge — The meal challenge scheduled for 4-6 days after the patient's last injection. The study team will insert an indwelling venous catheter into the participant's forearm for serial blood draws. Immediately prior to the meal, participants will consume 1500 mg of acetaminophen (off-label) to facilitate the analysis of gastric emptying. The participant will then begin the meal challenge by eating the test meal, a breakfast casserole, containing 33% of their current resting energy expenditure needs estimated by Mifflin-ST Jeor equation with a composition of 50% carbohydrate, 30% fat and 20% protein. Participants must completely consume the test meal within 25 minutes of initiating the meal. Participants will fill out behavioral questionnaires after consuming the test meal. After the 2-hour blood draw period, participants will be dismissed. Blood will be drawn prior to the meal and at 5, 10, 15, 30, 60, 90, and 120 minutes after initiating the meal.

SUMMARY:
This study aims to explore how anti-obesity medications (AOMs) like semaglutide and tirzepatide affect appetite and energy intake. Researchers will examine two groups: one just starting AOMs and another that has already achieved significant weight loss and maintained it. By conducting meal challenges at different stages of medication use, the study will assess feasibility of the methods and gather preliminary data to design a larger, future study.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females with a BMI of 30-45 kg/m2 (early group), or a BMI of 30-45 kg/m2 prior to weight loss achieved through medication (late group)
* Age, 25-60 years old
* Passing medical and physical screening, and analysis of blood and urine screening samples
* Anticipated to start or are already prescribed AOMs (semaglutide or tirzepatide)
* 6-months weight stable (early group) or 3 months weight stable at current weight (late group)
* Women of reproductive age must be using an effective form of contraception

Exclusion Criteria:

* Diagnosed with type 1 or 2 diabetes
* Smoker
* Previous surgical treatment or device-based therapy for obesity
* Chronic or acute pancreatitis
* Clinically significant gastric emptying abnormality
* Uncontrolled hypertension or hypo/hyperthyroidism
* Cardiovascular event 3 months within screening
* Acute or chronic hepatitis
* Inability to tolerate beef, eggs, and cheese
* Women who are pregnant
* Women who are nursing

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Potential participants are residents of the Denver metropolitan area who have either:
  1. Had or has obesity and experienced significant weight loss while taking semaglutide or tirzepatide, or
  2. Has obesity and has established agreements with their healthcare providers to begin treatment with semaglutide or tirzepatide.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Participant Recruitment | 6-10 weeks
  Number of participants recruited for the study.
Meal test tolerability | 6-10 weeks
  Number or participants able to tolerate and complete the test meal.
Rate of protocol completion | 6-10 weeks
  Percentage of participants enrolled that complete the protocol

SECONDARY OUTCOMES:
Change in peptide YY (pg/ml) | 6-10 weeks
Change in Glucagon Like Peptide-1 (pg/mL) | 6-10 weeks
Change in leptin (ng/mL) | 6-10 weeks
Change in insulin (uIU/mL) | 6-10 weeks
Change in Glucagon (pg/mL) | 6-10 weeks
Glucose-Dependent Insulinotropic Peptide (pg/mL) | 6-10 weeks
Change in Glucose (mg/dL) | 6-10 weeks
Change in triglycerides (mg/dL) | 6-10 weeks
Change in free fatty acids (uEq/L) | 6-10 weeks
Change in Total Cholesterol (mg/dL) | 6-10 weeks
Gastric emptying by acetaminophen | 6-10 weeks
  Peak acetaminophen concentration in blood
Eating Rate | 6-10 weeks
  Calories/minutes
Changes in subjective hunger by visual analog scale (VAS) | 6-10 weeks
  Line from 0: not hungry to 10: extremely hungry
Changes in subjective fullness by visual analog scale (VAS) | 6-10 weeks
  Line from 0: not full to 10: extremely full
Changes in perceived prospective food consumption by visual analog scale (VAS) | 6-10 weeks
  Line from 0: no desire to eat more to 10: I could eat a large amount.
Changes in subjective nausea by visual analog scale (VAS) | 6-10 weeks
  Line from 0: no nausea at all more to 10: worst nausea possible.
Disinhibition measured by TFEQ | 6-10 weeks
  Disinhibition

IPD SHARING:
Plan to Share IPD: No